CLINICAL TRIAL: NCT06020404
Title: Physiological Effects of Prone vs. sUpine Position on Lung Recruitability in infantS/Children With Acute Respiratory Distress Syndrome
Brief Title: Prone Position in infantS/Children With Acute Respiratory Distress Syndrome
Acronym: PULSAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5922
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-08

CONDITIONS: Prone Position; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: 2x2 cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Experimental): Eligible patients will undergo the experimental protocol.
  Interventions: Procedure: supine position; Procedure: prone position
- Patients (Experimental): Eligible patients will undergo the experimental protocol.
  Interventions: Procedure: supine position; Procedure: prone position

INTERVENTIONS:
Procedure: supine position — At the end of the PEEP trial (i.e. at PEEP 5 cmH2O), patients will lay in the supine position for 15 minutes arterial blood gases will be performed and then a one-breath derecruitment maneuver (5-second exhalation, respiratory rate < 8 bpm) from PEEP 5 cmH2O to 0 cmH2O will be conducted to assess baseline functional residual capacity (FRC), defined as the EELI measured at 0 PEEP.
Procedure: prone position — After the supine step, each enrolled patient will be placed in the prone position for 1 hour.
  For safety reasons, enteral feeding will be interrupted 30 minutes before prone positioning and re-established after the study ending.
  During pronation FiO2 will be increased up to 80% and then gradually decreased to the baseline value within the first 30 minutes of prone positioning. After 30 minutes of PEEP 12 cmH2O (provided that plateau and driving pressures did not exceed 30 cmH2O and 15 cmH2O, respectively) to stabilize lung volumes, the same measurements applied for the supine step will be performed. Any further modifications in the MV settings will be discouraged over the entire course of the study; nonetheless, if needed to achieve the SpO2 target, an increase in FiO2 will be allowed and recorded.
  In case of sudden worsening of the oxygenation impairment or haemodynamic, 100% FiO2 will be set, and the patient will be promptly positioned in the supine semi-recumbent position.

SUMMARY:
In adult patients with acute respiratory distress syndrome (ARDS), the beneficial effects of prone position (PP) have been well investigated and explored; it reduces intrapulmonary shunt (Qs/Qt) and enhances lung recruitment, modifying both lung ventilation (VA) and lung perfusion (Q) distribution, finally generating an improvement in VA/Q matching and reversing oxygenation impairment;it reduces right ventricular afterload, increase cardiac index in subjects with preload reserve and reverse acute cor pulmonale in severe ARDS patients, but in infants and children there is still a lack of clear evidence. Taken together, these effects explain why PP improves oxygenation, limits the occurrence of ventilator-induced lung injury and improves survival.

Prone position is simple to perform in infants and in some neonatal and pediatric intensive care units is already commonly accomplished. However, a detailed analysis of the respective effects of high PEEP and prone position is lacking in infants/children with ARDS, while these two tools may interfere and/or act coherently. A recent multicenter, retrospective analysis of patients with pediatric acute respiratory distress syndrome (PARDS) describes how patients managed with lower PEEP relative to FIO2 than recommended by the ARDSNet model had higher mortality, suggesting that future clinical trials targeting PEEP management in PARDS are needed. We designed a physiological study to investigate the physiological effects of prone positioning on lung recruitability in infants/children with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Each patient meeting inclusion criteria will be evaluated for the presence of the oxygenation criterion. After neuromuscular paralysis (or apnoeic ventilation as per PICU protocol), and endotracheal suctioning, eligible patients will be ventilated for 30 min with PEEP = 5 cmH2O in the semi-recumbent position, with a tidal volume limited to 6 mL/kg and a Plateau Pressure less than 30 cmH2O. FiO2 will be titrated to obtain and SpO2 >92 % and <98 %. Afterward, arterial blood gas analysis (ABG) will be performed to compute PaO2/FiO2 ratio to confirm the presence of the inclusion and the absence of exclusion criteria.Patients showing PaO2/FiO2 ≤ 200 mmHg will be enrolled. Eligible patients will undergo the following protocol:

* Verify the presence of airway closure with airway opening pressure (AOP) > PEEP5cmH2O;
* PEEP will be initially set at 12 cmH2O (providing that plateau and driving pressures do not exceed 30 cmH2O and 15 cmH2O, respectively) for 40 minutes to stabilize lung volumes; afterwards, respiratory mechanics will be assessed through standard occlusions and arterial blood gases will be analyzed. Subsequently, a 4-steps decremental PEEP trial (PEEP 12 to 10 to 8 to 5 cmH2O) will be conducted. Each PEEP step will last 8 minutes, and all other ventilator settings will remain unchanged throughout the procedure. At the end of each PEEP step respiratory mechanics will be assessed by the ventilator through 1-second end-inspiratory and end-expiratory holds: plateau pressure [Pplat] and total PEEP [PEEPtot] will be measured, and driving pressure [ΔP=Pplat-PEEPtot] and respiratory system compliance [Crs = VT/ΔP] will be assessed;
* End-expiratory lung impedance (EELI) will be measured by electrical impedance tomography (EIT)

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 < 200 in the supine position, with a standard PEEP of 5 cmH2O;
* PaCO2 <45mmHg;
* Absence of history of chronic respiratory disease or heart failure or congenital heart disease (Modified Ross heart failure classification for children < II);
* Not underweight infants/children defined as a low body mass index (BMI) for age;
* Absence of any contraindication to PP (Appendix 1);
* Written informed consent of both parents and the legal guardian.

Exclusion Criteria:

* Barotrauma;
* Less than 4 weeks of age (new-born physiology);
* Exacerbation of asthma;
* Chest trauma;
* Pulmonary oedema/haemorrhage;
* Severe Neutropenia (<500 WBC/mm3);
* Haemodynamic instability (Systolic blood pressure < 5th percentile or mean arterial pressure < 5th percentile adjusted by age);
* Lactic acidosis (lactate >5 mmol/L) and/or clinically diagnosed shock;
* Metabolic Acidosis (pH <7.30 with normal- or hypo-carbia);
* Chronic kidney failure requiring dialysis before PICU admission;
* Upper gastrointestinal bleeding.
* Refusal to sign written informed consent of both parents and the legal guardian.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
effect of prone positioning on lung recruitability | at the end of the supine and prone position
  PaO2/FiO2 ratio

SECONDARY OUTCOMES:
difference in gas exchanges | at the end of the supine and prone position
  PaO2/FiO2, PaCO2, PaO2
ventilatory ratio | at the end of the supine and prone position
  minute ventilation (ml/min) × PaCO2 (mmHg)]/(predicted body weight × 100 × 37.5)
global impedance-derived End-expiratory lung volume | at the end of the supine and prone position
  effects of prone position on End-expiratory lung volume, measured with electrical impedance tomography
regional impedance-derived End-expiratory lung volume | at the end of the supine and prone position
  effects of prone position on End-expiratory lung impedance in the four regions of the lungs (ventral, mid-ventral, mid-dorsal, dorsal), measured with electrical impedance tomography
tidal volume distribution | at the end of the supine and prone position
  effect of prone position on % tidal volume distribution in the four regions of the lung (ventral, mid-ventral, mid-dorsal, dorsal), explored with electrical impedance tomography
global impedance-derived lung dynamic strain | at the end of the supine and prone position
  change in impedance due to tidal volume / end expiratory lung impedance, both measured with electrical impedance tomography
regional impedance-derived lung dynamic strain | at the end of the supine and prone position
  change in impedance due to tidal volume / end expiratory lung impedance in the four regions of the lungs (ventral, mid-ventral, mid-dorsal, dorsal), measured with electrical impedance tomography
number of displacements of the endotracheal tube during prone position | 2 hours
  safety endpoint
number of oxygen desaturations during prone position | 2 hours
  safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Giorgio Conti, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Pelosi P, Tubiolo D, Mascheroni D, Vicardi P, Crotti S, Valenza F, Gattinoni L. Effects of the prone position on respiratory mechanics and gas exchange during acute lung injury. Am J Respir Crit Care Med. 1998 Feb;157(2):387-93. doi: 10.1164/ajrccm.157.2.97-04023. PMID 9476848
- [Result] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Result] Curley MA, Hibberd PL, Fineman LD, Wypij D, Shih MC, Thompson JE, Grant MJ, Barr FE, Cvijanovich NZ, Sorce L, Luckett PM, Matthay MA, Arnold JH. Effect of prone positioning on clinical outcomes in children with acute lung injury: a randomized controlled trial. JAMA. 2005 Jul 13;294(2):229-37. doi: 10.1001/jama.294.2.229. PMID 16014597
- [Result] Lupton-Smith A, Argent A, Rimensberger P, Frerichs I, Morrow B. Prone Positioning Improves Ventilation Homogeneity in Children With Acute Respiratory Distress Syndrome. Pediatr Crit Care Med. 2017 May;18(5):e229-e234. doi: 10.1097/PCC.0000000000001145. PMID 28328787
- [Result] Bhandari AP, Nnate DA, Vasanthan L, Konstantinidis M, Thompson J. Positioning for acute respiratory distress in hospitalised infants and children. Cochrane Database Syst Rev. 2022 Jun 6;6(6):CD003645. doi: 10.1002/14651858.CD003645.pub4. PMID 35661343
- [Result] Fineman LD, LaBrecque MA, Shih MC, Curley MA. Prone positioning can be safely performed in critically ill infants and children. Pediatr Crit Care Med. 2006 Sep;7(5):413-22. doi: 10.1097/01.PCC.0000235263.86365.B3. PMID 16885792
- [Result] Khemani RG, Parvathaneni K, Yehya N, Bhalla AK, Thomas NJ, Newth CJL. Positive End-Expiratory Pressure Lower Than the ARDS Network Protocol Is Associated with Higher Pediatric Acute Respiratory Distress Syndrome Mortality. Am J Respir Crit Care Med. 2018 Jul 1;198(1):77-89. doi: 10.1164/rccm.201707-1404OC. PMID 29373802
- [Result] Sinha P, Calfee CS, Beitler JR, Soni N, Ho K, Matthay MA, Kallet RH. Physiologic Analysis and Clinical Performance of the Ventilatory Ratio in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2019 Feb 1;199(3):333-341. doi: 10.1164/rccm.201804-0692OC. PMID 30211618
- [Result] Menga LS, Delle Cese L, Rosa T, Cesarano M, Scarascia R, Michi T, Biasucci DG, Ruggiero E, Dell'Anna AM, Cutuli SL, Tanzarella ES, Pintaudi G, De Pascale G, Sandroni C, Maggiore SM, Grieco DL, Antonelli M. Respective Effects of Helmet Pressure Support, Continuous Positive Airway Pressure, and Nasal High-Flow in Hypoxemic Respiratory Failure: A Randomized Crossover Clinical Trial. Am J Respir Crit Care Med. 2023 May 15;207(10):1310-1323. doi: 10.1164/rccm.202204-0629OC. PMID 36378814
- [Result] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Result] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Result] Bachmann MC, Morais C, Bugedo G, Bruhn A, Morales A, Borges JB, Costa E, Retamal J. Electrical impedance tomography in acute respiratory distress syndrome. Crit Care. 2018 Oct 25;22(1):263. doi: 10.1186/s13054-018-2195-6. PMID 30360753
- [Result] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Result] Baudin F, Emeriaud G, Essouri S, Beck J, Portefaix A, Javouhey E, Guerin C. Physiological Effect of Prone Position in Children with Severe Bronchiolitis: A Randomized Cross-Over Study (BRONCHIO-DV). J Pediatr. 2019 Feb;205:112-119.e4. doi: 10.1016/j.jpeds.2018.09.066. Epub 2018 Nov 14. PMID 30448014